CLINICAL TRIAL: NCT02479568
Title: Randomized, Parallel and Double Blind Placebo-controlled Study for the Evaluation of Both Acute and Chronic Role of Hesperidin Consumption in 100% Orange Juice
Brief Title: Beneficial Impact of Orange Juice Consumption on Risk Factors Associated With Cardiovascular Diseases
Acronym: CITRUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: Florida Department of Citrus (Other); Technological Centre of Nutrition and Health (Other); Hospital Universitari Sant Joan de Reus (Other); University Rovira i Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CITRUS 14-12
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Risk Factors
Keywords: Cardiovascular disease; biomarkers; transcriptomics; orange juice; hesperidin; systolic blood pressure; metabolomics; cardiovascular risk factor
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Control drink (placebo)
  Interventions: Dietary Supplement: Control
- Natural Florida orange juice (Experimental): 100% Florida orange juice (OJ) (natural content of hesperidin)
  Interventions: Dietary Supplement: 100% Florida OJ
- Enriched Florida orange juice (Experimental): 100% Florida orange juice (OJ) (enriched hesperidin content)
  Interventions: Dietary Supplement: 100% Florida OJ-enriched

INTERVENTIONS:
Dietary Supplement: Control — 500 mL (250 mL; 2 times/day) of placebo drink for 12 weeks
  Arms: Control
Dietary Supplement: 100% Florida OJ — 500 mL (250 mL; 2 times/day) of 100% Florida OJ for 12 weeks
  Arms: Natural Florida orange juice
Dietary Supplement: 100% Florida OJ-enriched — 500 mL (250 mL; 2 times/day) of 100% Florida OJ-enriched for 12 weeks
  Arms: Enriched Florida orange juice

SUMMARY:
The primary aim is to examine both the acute and chronic effects of hesperidin consumption from 100% Florida orange juice in various doses on functional and systemic markers associated with cardiovascular disease (CVD) risks.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of different doses of hesperidin in 100% Florida orange juice (OJ) when regularly or postprandially consumed on cardiovascular risk markers; in addition, the plausible role and mechanism of the hesperidin will be investigated.

The sample size was calculated using a previously available bibliography using systolic blood pressure (SBP) as the primary outcome measure. A total of 84 subjects per study product group were needed, assuming variance components of approximately 20.0, to detect differences between the three groups (control, orange juice and hesperidin-enriched orange juice (10 mm Hg)) with a bilateral significance level of α=0.05 and a power of 80 %.

The sample size was computed to be sufficient to detect differences between treatment groups regarding the evolution in time of SBP levels. Justification of chosen sample size is based on the clinically meaningful difference assigned to δ=10.0 mm Hg, which is equivalent to a difference of approximately 7.4 % in patients with baseline SBP levels of approximately 135 mm Hg. Thus, a sample of 252 participants can be used for the chronic three arm parallel trial design (84 subjects/arm) and will allow us to detect small but clinically relevant differences between the three groups with statistical robustness and direct interpretation in terms of the chronic treatment effect.

To the acute postprandial tests, the investigators have chosen n=20 subjects per arm according to the most studies that have addressed the metabolic effects of a postprandial intervention have been performed using a very similar number of subjects with statistically good quality results.

The statistical analysis will follow the principles specified in the guidelines of the ICHE9 and CPMP/EWP/908/99 ICHE9 Points to Consider on Multiplicity Issues in Clinical Trials.

The continuous efficacy variables will be analyzed by an ANCOVA (analysis of covariance) with the baseline value as a covariate.

The efficacy outcomes will be determined using the absolute values and absolute differences from the baseline. The efficacy analysis will be performed using the Available Data Only approach. In addition, the analysis of the primary efficacy variable will be performed with the Baseline Observation Carried Forward approach.

A suitable hypothesis test will be applied to the rest of the variables according to the nature of each variable, such as the Fisher exact test for categorical variables, Student's T-test for continuous variables and Mann-Whitney U test for ordinal scale variables.

The statistical tests will be applied with an α=0.05 two-sided significance level. Post-hoc analyses and comparisons between pairs of groups will be done as for exploratory purposes.

In addition, the statistical plan will be transferred to the application form of the electronic data collection report (e-CDR), which allows the improvement of data management, diminishes human errors (according threshold values of each outcome) and, overall, guarantees the maximum exploitation of human data in the context of statistical analysis.

ELIGIBILITY:
Inclusion criteria

* Men or women 18-65 years old
* No evidence of chronic disease
* No familial CVD history
* Written informed consent provided before the initial screening visit.
* Blood pressure (with no drug intervention) >120 mm Hg systolic blood pressure ≤ 159 mmHg

Exclusion criteria

* Body mass index (BMI) ≥ 35 kg/m2
* Glucose >125 mg/dl
* Systolic blood pressure ≥ 160 mm Hg and diastolic blood pressure >100 mm Hg or taking antihypertensive medications
* Total cholesterol >240 mg/dl
* LDL-cholesterol >160 md/dl
* TAG >350
* Smoking
* Pregnant or intending to become pregnant
* Use of medications, antioxidants, or vitamin supplements
* Chronic alcoholism
* Intense physical activity (5h/week)
* Intestinal disorders
* Following of a vegetarian diet
* Anemia (hemoglobin ≤13 g/dL in men and ≤12 g/dL in women)
* Current or past participation in a clinical trial or consumption of a research product in the 30 days prior to inclusion in the study
* Failure to follow the study guidelines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-01-12; Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Every 2 weeks for a total of 12 weeks.
  During each visit, SBP will be measured after 5 min in a seated position in a comfortable room by the physician. The measurement will be taken in duplicate at 1-min intervals using an automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain), and the average of the two measurements will be calculated.

SECONDARY OUTCOMES:
Diastolic Blood Pressure | Every 2 weeks for a total of 12 weeks.
  During each visit, diastolic BP will be measured after 5 min in a seated position in a comfortable room by the physician. The measurement will be taken in duplicate at 1-min intervals using an automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain), and the average of the two measurements will be calculated.
Ischemic reactive hyperemia (IRH) | Every 4 weeks for a total of 12 weeks
  The endothelial-dependent vasomotor functions will be measured as IRH by a Laser-Doppler linear Periflux 5000 flowmeter (Perimed AB, Järfälla, Stockholm, Sweden)
Platelet aggregation | Every 4 weeks for a total of 12 weeks
  Multiplate analyzer, Roche
Homocysteine | Every 4 weeks for a total of 12 weeks
  Homocysteine concentrations will be measured by liquid chromatography-mass spectrometry (LC-MS/MS)
C-reactive protein (inflammatory marker) | Every 4 weeks for a total of 12 weeks
  High sensitivity C-reactive protein (hsCRP) by standardized methods in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain)
oxidized LDL (as oxidative stress biomarker) | Every 4 weeks for a total of 12 weeks
  Mercodia Oxidized LDL ELISA kit will be used to measure the oxidized LDL (mU/L).

OTHER OUTCOMES:
Transcriptomics | At week 0 (V1) and 12 week (V7).
  Plasma collected at 0 h (V1 and V7) of 20 samples each arm (volunteers in the postprandial study). These cells will be used to perform transcriptomics analysis to detect whole gene expression changes due to the chronic consumption of two doses of hesperidin in 100% Florida orange juice.
Non-targeted Metabolomics | At week 0 (V1) and 12 week (V7).
  Plasma collected at 0 h (V1 and V7) of 20 samples each arm (volunteers in the postprandial study) will be used to perform non-targeted metabolomics by Nuclear Magnetic Response Spectroscopy (NMR) to detect metabolomic profile changes due to the chronic consumption of two doses of hesperidin in 100% Florida orange juice

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà Alberich, Prof, MD, Principal Investigator — • University Rovira i Virgili / Hospital Universitari Sant Joan de Reus
Locations (1):
- Technological Centre of Nutrition and Health (CTNS), Reus, Tarragona, Spain

REFERENCES:
- See also: Technological Centre of Nutrition and Health — http://www.ctns.cat/en
- See also: Florida Department of Citrus — http://fdocgrower.com/